CLINICAL TRIAL: NCT02885935
Title: Dairy Macronutrient Effects on the Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: Dairy Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 138447
Record Dates: First submitted 2016-08-24; First posted 2016-09-01 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2016-08

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Recommended protein intake (Experimental): Subjects consumed diets with a macronutrient distribution of 10% protein, 55% carbohydrates, and 35% fat for 4 weeks.
  Interventions: Other: Recommended protein intake
- Elevated protein intake (Experimental): Subjects consumed diets with a macronutrient distribution of 20% protein, 45% carbohydrates and 35% fat for 4 weeks.
  Interventions: Other: Elevated protein intake

INTERVENTIONS:
Other: Recommended protein intake — Recommended protein intake diet contained 10% protein, 55% carbohydrate,and 35 % fat.
  Arms: Recommended protein intake
Other: Elevated protein intake — Recommended protein intake diet contained 20% protein, 45% carbohydrate,and 35 % fat.
  Arms: Elevated protein intake

SUMMARY:
The investigators examined the effects of 4-week dietary protein intake in mixed meals at two levels of protein amount on whole body glucose metabolisms in older adults with metabolic syndrome.

DETAILED DESCRIPTION:
The investigators investigated changes in insulin sensitivity before and after 4 weeks of dietary intervention and control in subjects with metabolic syndrome. Two groups of subjects were studied before and after a weight maintenance diet. Group 1 was fed a common American diet with a macronutrient distribution of 10% protein, 55% carbohydrates, and 35% fat. Group 2 consumed a higher protein diet (20%; 1.4 g/kg/d of protein). Carbohydrate intake was lower in Group 2 (45%), with fat intake (largely derived from dairy sources) similar between groups. Glucose utilization and endogenous glucose production were determined during an oral glucose tolerance test (OGTT) with a novel double-tracer approach. The secondary aim was to determine the effect of a diet high in dairy consumption on blood lipid profiles. The investigators measured blood lipids before and after dietary intervention in each group.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, ages 45-75 years AND
* BMI greater than 30 kg/m2 AND
* Two of the following conditions:

  * Plasma triglycerides > 130 mg/dl
  * HDL < 40 mg/dl in men or 50 mg/dl in women
  * elevated screening blood pressure (systolic > 140 or diastolic >90 mm Hg) or taking medication for hypertension
  * fasting plasma glucose > 100mg/dl

Exclusion Criteria:

* Hemoglobin A1c > 7.5
* History of malignancy in the 6 months prior to enrollment
* History of lactose intolerance or dairy allergy
* History of gastrointestinal bypass surgery (Lapband, etc)
* History of a chronic inflammatory condition or disease (Lupus, HIV/AIDS, etc)
* Subjects who do not or will not eat animal proteins
* Subjects who cannot refrain from consuming protein or amino acid supplements during their participation in this study
* Subjects who use insulin to control their blood sugar
* Subjects whose physician will not allow suspension of oral diabetes medications for the duration of the study (~5 weeks)
* Concomitant use of corticosteroids (ingestion, injection or transdermal)
* Any other disease or condition that would place the subject at increased risk of harm if they were to participate, at the discretion of the study physician

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-04; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Changes in rate of glucose disappearance | Change from baseline and after 4weeks of dietary intervention
  Rate of glucose disappearance from plasma to body tissues is a measure of whole body insulin sensitivity

REFERENCES:
- [Derived] Kim IY, Schutzler SE, Azhar G, Wolfe RR, Ferrando AA, Coker RH. Short term elevation in dietary protein intake does not worsen insulin resistance or lipids in older adults with metabolic syndrome: a randomized-controlled trial. BMC Nutr. 2017;3:33. doi: 10.1186/s40795-017-0152-4. Epub 2017 Apr 17. PMID 28713581